CLINICAL TRIAL: NCT01299831
Title: THE RELATIONSHIP BETWEEN BODY COMPOSITION AND GROWTH HORMONE, SIRT SIGNALING, PROTEIN TURNOVER AND INSULIN SENSITIVITY. Studies of Signaling Pathways in Fat and Muscle, and Turnover of Protein, Sugar and Fat After Stimulation With Growth Hormone and During Fasting in Lean and Obese Subjects
Brief Title: The Relationship Between Body Composition and Growth Hormone, SIRT Signaling, Protein Turnover and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M-2010082
Record Dates: First submitted 2011-01-21; First posted 2011-02-18 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — Growth Hormone; acipimox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 72 hour fast (Experimental)
  Interventions: Behavioral: 72 hour fast
- 12 hours fast (Experimental)
  Interventions: Behavioral: control, 12 hour fast
- 12 hour fast, growth hormone bolus (Experimental)
  Interventions: Drug: Growth hormone
- 72 hour fast, inhibition of lipolysis (Experimental)
  Interventions: Drug: Olbetam

INTERVENTIONS:
Behavioral: 72 hour fast — The participants will be fasting 72 hours prior to the start of the study day, drinking water is allowed.
  Arms: 72 hour fast
Behavioral: control, 12 hour fast — The 12 hour fast will be used as a basic metabolic control
  Arms: 12 hours fast
Drug: Growth hormone — Genotropin bolus(0,005 mg/kg over 20 min.) will be administered at the beginning of the study day after a 12 hour fast.
  Arms: 12 hour fast, growth hormone bolus
Drug: Olbetam — The participants will be fasting 72 hours prior to the start of the study day, drinking water is allowed.
  During the last 12 hours of fasting and the study day lipolysis will be inhibited with one tablet of olbetam 250 mg every 4 hours.
  Arms: 72 hour fast, inhibition of lipolysis

SUMMARY:
The purpose of this study is to investigate signaling pathways in fat and muscle, as well as turnover of protein, sugar and fat after stimulation with growth hormone and during fasting in lean and obese subjects. This will help clarify differences in the human metabolism between lean and obese subject and provide us with a better understanding of the molecular mechanisms regulating the basic metabolism during prolonged fasting.

DETAILED DESCRIPTION:
In an evolutionary context, it is likely that "inherited" obesity provides a survival advantage when there are shortages of food, but also increases the risk of lifestyle diseases in times of prosperity. This may explain the high incidence of obesity, diabetes and cardiovascular disease in the western world today. Obese individuals have high levels of free fatty acids (FFAs) in the blood and FFAs are both protein sparing (giving an evolutionary survival advantage) but also cause increased insulin resistance (which increases the risk of diabetes and cardiovascular disease). Obesity also leads to low growth hormone (GH)-levels, whereas fasting is accompanied by high GH- and FFA-levels and increased IGF-I mRNA in muscle. It is likely that obese individuals are more capable of fasting than lean individuals and will lose less protein during fasting, have increased activation of GH signaling and altered activation of other signaling proteins. And obese individuals are likely to be more sensitive to growth hormone than lean individuals based on FFA-responses, intracellular signaling, protein loss and insulin sensitivity.

We would like to test 3 hypotheses: (1) Obese individuals are more capable of fasting than lean individuals and will lose less protein during fasting (2) Activation of lipolysis is an important prerequisite for limiting protein loss during fasting in both slim as obese individuals. (3) Obese individuals are more sensitive to growth hormone than lean individuals based on FFA responses and activation of intracellular signals. The hypotheses are tested in 8 lean and 8 obese healthy young men, who are studied 4 times: (i) after 12 hours of fasting (ii) after 72 hours of fasting (iii) after GH-bolus (0.005 mg/kg over 20 min.) and (iv) after 72 hours of fasting with inhibition of fat metabolism (tablet acipimox 250 mg every 4 hours) during the last 12 hours of fasting and during the study period.

Each study period consists of a 4-hour basal period and a 2 hour hyperinsulinemic euglycemic clamp (30 mU/m2/min). Muscle- and fat-biopsies are taken and analyzed for enzyme expression and activation of various signaling pathways. The study subjects are given glucose-, amino acid-, urea- and palmitate-tracers and specific hormones and metabolites are measured for assessment of underlying molecular mechanisms regulating the basic human energy metabolism.

ELIGIBILITY:
Inclusion Criteria:

* healthy lean (BMI19-25) and healthy obese (BMI 32-40) men
* written consent before study start

Exclusion Criteria:

* known medical conditions
* any medication

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Measurements of changes in metabolism | 6 hours
  Measurements of the switch to lipid metabolism during fasting in lean and obese human subjects.

SECONDARY OUTCOMES:
Signaling pathways in muscle and fat tissue involved in regulation of metabolism | 6 hours
  Protein and gene-exspression, phosphorylation and acetylation of specific proteins involved in lipid-, glucose and protein metabolism.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of medical endocrinology, University Hospital of Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Hogild ML, Bak AM, Pedersen SB, Rungby J, Frystyk J, Moller N, Jessen N, Jorgensen JOL. Growth hormone signaling and action in obese versus lean human subjects. Am J Physiol Endocrinol Metab. 2019 Feb 1;316(2):E333-E344. doi: 10.1152/ajpendo.00431.2018. Epub 2018 Dec 21. PMID 30576246